CLINICAL TRIAL: NCT00478114
Title: An Open-label, Non-comparative, Treatment Protocol for the Use of BAY 43-9006 (Sorafenib) in Patients With Advanced Renal Cell Carcinoma
Brief Title: Efficacy and Safety of Sorafenib in Advanced Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12750
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Sorafenib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sorafenib
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — sorafenib in the patients with advanced Renal Cell Carcinoma
  Other Names: nexavar

SUMMARY:
This is the early access programme (EAP) of sorafenib in the indication of advanced renal cell carcinoma (RCC). The study is to evaluate the efficacy and safety of sorafenib in patients with advanced RCC.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounts for approximately 3 % of all cancers. RCC can be cured if diagnosed and treated when still localized to the kidney or immediate surrounding tissues. Since most of the RCC tumours are diagnosed when still localized, approximately 40 % of all patients survive 5 years. The median survival of Stage IV RCC after diagnosis is 8 to 12 months and the 5-year survival is less than 10 %. Surgery has been the primary therapy for RCC for more than a century. Until recently, metastatic disease has been refractory to any systemic therapy. Despite recent advances in immunotherapy (e.g. Interferon and Interleukin-2), the response rates remain low (15 %) and few patients experience durable remission. Surgical and radiation therapies for Stage IV disease are generally limited to palliation of symptoms. For the majority of patients, metastatic RCC is incurable and patients should be considered candidates for clinical trials when appropriate. In summary, the available therapies for advanced unresectable and/or metastatic RCC have limited clinical values, with response rates ranging from 6-20 % and little impact on the natural history of the disease. Furthermore, the toxicities associated with these agents can be severe, requiring careful patient selection, and this dramatically decreases the number of patients who may benefit from therapy. Advanced RCC remains incurable and the need for more effective therapies is high.

This is a non-randomized, open-label treatment protocol for patients with advanced RCC. Patients will be treated with 400 mg oral sorafenib twice a day on a continuous. Patients in this protocol may continue to be treated with sorafenib as a single agent until any of the following criteria for drug or protocol discontinuation is reached:

1. Progression of disease.
2. The patient is unlikely to benefit from further treatment with sorafenib as judged by the Investigator.
3. Intolerable toxicity of the drug.
4. Withdrawal of consent for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to receiving sorafenib.
2. At least 18 years of age.
3. Advanced Renal Cell Carcinoma.
4. A patient who has received prior systemic and local therapies, must have completely recovered from acute toxicity (i.e. resolved back to CTC-AE Grade 1 or less).
5. For patients, who have had major surgery or injury, the wound must be completely healed prior to receiving sorafenib treatment (4 weeks).
6. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Men must use adequate birth control for at least 3 months after the last administration of sorafenib. Should a woman become pregnant while participating or while the partner of a patient is participating in the study, they should inform their treating physician immediately.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Patients with metastatic brain or meningeal tumours.
3. Cardiac disease: greater than NYHA functional class II; unstable CAD; MI within the last 6 months.
4. HIV infection or chronic hepatitis B or C; patients with Child-Pugh class C hepatic impairment.
5. Patients with severe renal impairment (calculated creatinine clearance of < 30 ml/min) or who require dialysis.
6. Patients with active uncontrolled hypertension.
7. Patients with recent or active bleeding diathesis.
8. Patients with any medical condition which could jeopardize their safety while taking an investigational drug.
9. Excluded therapies or medications, previous and concomitant:

   * Bone marrow transplant or stem cell rescue within 4 months of study entry.
   * Anticipation of the need for major surgery during the course of the study.
   * CYP 3A4 inducers (e.g. rifampicin, St. John's Wort [Hypericum perforatum], phenytoin, phenobarbital and dexamethasone).
10. Any investigational therapy while on this protocol or within 30 days prior to their first dose of sorafenib.

    * Any drugs (licensed or investigational) that targets angiogenesis, especially VEGF or VEGF-Receptors (e.g. bevacizumab).
    * Any drug (licensed or investigational) that targets Ras-pathway or EGFR.
    * Biological response modifiers, such as G-CSF or GM-CSF, within 3 weeks prior to study entry or during study (G-CSF and other hematopoietic growth factors may only be used in the management of acute toxicity such as febrile neutropenia, when medically indicated or at the discretion of the Investigator).
    * Use of Megestrol-acetate and medroxyprogesterone.
    * Patients taking narrow therapeutic index medications will be monitored closely.
    * These include warfarin, phenytoin, quinidine, carbamazepine, phenobarbital, cyclosporine and digoxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (time to progression and progression free survival) of sorafenib in patients with advanced RCC | two years

SECONDARY OUTCOMES:
To evaluate the safety (all drug-related adverse events, all adverse events NCI CTCAE 3.0 Grade 3 or higher) of sorafenib in patients with advanced RCC | two years

CONTACTS AND LOCATIONS:
Overall Officials: Vichien Srimuninnimit, Ass.Prof., Principal Investigator — Siriraj Hospital, Bangkok, Thailand
Locations (1):
- Siriraj Hospital, Department of Medicine, Bangkoknoi, Bangkok, Thailand